CLINICAL TRIAL: NCT00873379
Title: Melatonin Supplementation for Delirium Prevention in Acutely Hospitalized Elderly: a Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Melatonin Supplementation for Delirium Prevention in Acutely Hospitalized Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Chris brymer, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-07-314; 13426
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- melatonin (Active Comparator): .5 mg (one half of a 1 mg tablet of GNC rapid dissolving Melatonin, natural product number (NPN) 80001380)
  Interventions: Dietary Supplement: melatonin
- placebo (Placebo Comparator): half a white placebo tablet
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: melatonin — one half of a 1 mg tablet of GNC rapid dissolving Melatonin, NPN (natural product number) 80001380, available over the counter in Canada
  Arms: melatonin
Dietary Supplement: placebo — half a white placebo tablet
  Arms: placebo

SUMMARY:
122 people over 70 who were admitted to hospital were enrolled to the study. Half got .5 mg a night of melatonin, half got a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 admitted through the emergency department to an internal medicine service in London, Ontario, Canada.

Exclusion Criteria:

* Life expectancy less than 24 hours,
* Unable to communicate in English,
* Unable to take oral medications,
* Intracranial bleed or known seizure disorder,
* Markedly sub or supra-therapeutic INR while on warfarin, OR
* A known allergy to study tablet ingredients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
delirious using confusion assessment method (CAM) | days

SECONDARY OUTCOMES:
MDAS (memorial delirium assessment scale) | days

CONTACTS AND LOCATIONS:
Overall Officials: Chris Brymer, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada